CLINICAL TRIAL: NCT00414947
Title: A Single Center, Randomized, Open-Label, Crossover, Single Oral Dose Study to Assess the Bioequivalence of LAF237 Tablet Manufactured by Beijing Novartis Pharma Ltd. to Imported LAF237 Tablet in Chinese Healthy Subjects
Brief Title: Bioequivalence of Vildagliptin Tablet Manufactured in China Compared to Imported Vildagliptin Tablet in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A2111
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Bioequivalence; safety; LAF237; vildagliptin; Chinese; healthy subjects
MeSH Terms: interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

INTERVENTIONS:
Drug: Vildagliptin (LAF237)

SUMMARY:
This study will evaluate the bioequivalence as well as rate and extent of absorption of vildagliptin tablet manufactured by Beijing Novartis Pharma Ltd. compared to the imported vildagliptin tablet in Chinese healthy volunteers.

This trial is not recruiting patients in the United States,

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male subjects age 18 to 40 years of age included
* In good health
* Male subjects using a double-barrier local contraception for the entire duration of the study up to study completion visit and refraining from fathering a child in the three months following last study drug administration.
* Body mass index within the range of 19 to 24 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Smokers
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Paracetamol is acceptable.
* Participation in any clinical investigation within 4 weeks prior to dosing.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities.
* History of:

  * Fainting, low blood pressure when standing, irregular heartbeats,
  * Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated),
  * Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis)
  * Known hypersensitivity to the study drug or similar drugs
  * Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or jeopardize participation in the study.
  * Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* Drug or alcohol abuse within the 12 months prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-12

PRIMARY OUTCOMES:
Rate and extent of absorption of vildagliptin tablet manufactured by Beijing Novartis Pharma Ltd. to imported vildagliptin tablet in Chinese healthy subjects

SECONDARY OUTCOMES:
Safety and tolerability of vildagliptin tablet after a 50 mg single dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Beijing, China